CLINICAL TRIAL: NCT05866094
Title: Feasibility Study of an Intervention to Provide Nutritional Care for People Living With Dementia at Home
Brief Title: nuTritiOn and deMentia AT hOme (TOMATO)
Acronym: TOMATO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bournemouth University (Other)
Collaborators: Leeds Beckett University (Other); University of Leeds (Other); University of Exeter (Other); Homecare Association (Unknown); Leeds Comunity Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2223/TOMATO/ IRAS1
Record Dates: First submitted 2023-04-24; First posted 2023-05-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Dementia; Undernutrition
Keywords: Dementia; Alzheimer's disease; Malnutrition; Undernutrition; Nutritional Care; Food; Eating; Drinking; Community; Home Care; Older adults; Ageing
MeSH Terms: conditions — Dementia; Malnutrition; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Participants: People with dementia, their relatives, and home care workers
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutrition Intervention (Experimental): Intervention Feasibility Testing (11-months, Phase 2)
  Interventions: Behavioral: Nutritional Intervention

INTERVENTIONS:
Behavioral: Nutritional Intervention — Nutrition training will be provided to home care staff to deliver the intervention via the participating Home Care Providers from two localities (South and North of England).
  This phase will involve identification of people with dementia on their caseload, preliminary assessment of potential impact via collection of quantitative data at baseline (pre-intervention), and at 4 months follow-up (4 months after the first visit by trained home care workers, following baseline).
  A process evaluation will be conducted to gather data on intervention fidelity and implementation (quantitative and qualitative).

SUMMARY:
The purpose of this study is to refine, implement and assess the acceptability and feasibility of an existing nutrition intervention applied to people living with dementia receiving home care.

DETAILED DESCRIPTION:
In the United Kingdom, two-thirds of people with dementia live at home and rely on family and friends to support with eating and drinking. Making sure people eat and drink well when they have dementia can be difficult as dementia progresses. Many with dementia are therefore at risk of being undernourished. This can be caused by poor appetite as well as eating and swallowing problems. Being undernourished can lead to poorer health and quality of life for people with dementia (and their carers), increased hospital admissions and health care use costing around £23.5 billion in terms of health and social care expenditure.

Home care workers provide care for people with dementia more frequently and for longer than healthcare professionals. Existing research and our engagement work indicate home care workers are well positioned to assess nutritional status and intervene early, but currently lack training, access to resources and support from NHS services. A more pro-active and wide-ranging approach to nutritional assessment and management is needed targeting interventions at home care workers and family carer dyads, with input from appropriate healthcare professionals.

As a collaborative project, the TOMATO study aims to work together with home care workers, people with dementia, and family carers to adapt a nutrition intervention (initially developed for care home) to support people living with dementia at home with eating and drinking. The intervention includes training programme, toolkit with video, workbook and guides for staff and family carers, and resources and leaflets.

This study will take place in Dorset, Midlands and West Yorkshire in two phases.

Phase 1: The first phase involves adapting the existing nutrition intervention by getting feedback from people with dementia, family carers, home care staff and nutrition experts through semi-structured interviews.

Phase 2: The second phase involves training home care workers to deliver the adapted approach to people with dementia and family carers (up to 32 participant dyads) in receipt of care at home. Information about food intake, weight, practicality, and costs of the approach will be gathered. Semi-structured interviews will also be conducted with participants living with dementia, their family carers, and home care managers to get their feedback on the approach.

If feasible and acceptable (based on progression criteria), findings will inform the design of future trial (effectiveness/implementation research).

The TOMATO patient and public involvement group which consist of family carers, people with dementia and home care workers will provide input throughout the study duration (including project design, delivery, analysis, reporting and dissemination of the findings).

ELIGIBILITY:
Participants: People with dementia, their relatives, and home care workers

Inclusion Criteria:

People with Dementia

* formal diagnosis or functional symptoms associated with probable dementia (assessed by a senior home care worker using the FAST).
* have family member/friend providing care/support and resident in the same house as the person with dementia or living close by.
* be currently or have recently (in last 6-months) been at risk of/experienced malnutrition in receipt of home care services.

  - For interviews, people with dementia will
* be able to communicate fluently enough in English or provide informed consent with the assistance of a translator or family member to participate.
* be able to recall their experiences of malnutrition and carer/home care worker responses well enough to discuss.

Carers and Home Care Workers

* currently or have recently (in last 6-months) provided care for someone with dementia at risk of/experiencing malnutrition.
* able to communicate fluently enough in English or provide informed consent with the assistance of a translator or family member to participate.

Exclusion Criteria:

People with Dementia

* Who are at end of life or on an end-of-life care pathway.
* Permanently cared for in bed.
* Do not have an informal caregiver.
* having specialist nutritional support e.g., feeding via tube.

Carers and Home Care Workers

* have not recently (in last 6-months) provided care for someone with dementia at risk of/experiencing malnutrition.
* not able to communicate fluently enough in English or provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Nutrition Intervention Refinement | Phase 1 - 4 Months
  Exploring the perspective of participants in phase 1 via semi-structured in-depth interviews (people with dementia, their family carers, and home care staff).
  • Qualitative analysis will be carried out to understand more about how nutritional care is currently provided for people with dementia at home and how our existing nutrition intervention can be adapted for home care.
Intervention Feasibility and Acceptability Testing | Phase 2 - 11 Months
  1. Recruitment:
     Percentage of participants recruited from participating home care provider.
  2. Attrition rate:
     Percentage of participants who drop out of the study before completion.
  3. Qualitative analysis of the feasibility and acceptability of the adapted intervention from the perspective of people with dementia, their family carers, and home care staff and healthcare professionals.

SECONDARY OUTCOMES:
Nutritional status | Phase 2 - 11 Months
  Preliminary assessment at baseline and 4 months follow up:
  a. Nutritional status
  - Body Mass Index (BMI): Body weight (kg) and height (m2) will be combined to determine BMI (weight (kg) / height (m2)).
  BMI of < 20 kg/m2 will be an indicator of undernutrition.
Health-related quality of life | Phase 2 - 11 Months
  Preliminary assessment at baseline and 4 months follow up:
  b. Health-related quality of life for people with dementia and carers will be measured using
  * EuroQol 5-Dimension 5-Level (EQ-5D-5L) with a scale from 0 to 100; higher scores indicate better quality of life.
  * Dementia Quality of Life questionnaire (DEMQoL) and DEMQoL-Proxy; 4-point scale, higher scores indicate better quality of life.
Functional status | Phase 2 - 11 Months
  Preliminary assessment at baseline and 4 months follow up:
  c. Functional status
  * Functional status (Deterioration in Daily Living Activities in Dementia) using Modified Barthel Index measures; 2-point scale rating with 0 to 20 points. Higher score indicates greater independence.
  * Functioning status using Lawton-Brody Instrumental Activities of Daily Living Scale; 4-point scale. Higher scores indicate greater independence and better functional ability.
Carer burden | Phase 2 - 11 Months
  d. Carer burden using Zarit Burden Interview; 0 to 88 points; higher scores indicate severe burden.
Process Evaluation | 11 Months [Phase 2
  Process Evaluation at 4 months: a process evaluation to gather data on intervention fidelity and implementation.
  1. Semi-structured interviews conducted individually, in pairs or small groups with participant dyads (family carers will be given the option to have a separate interview), home care workers and managers from the participating regions.
  2. Associated costs variables to deliver the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Murphy, PhD, Principal Investigator — Bournemouth University
Locations (5):
- United Kingdom (5):
  - Participating Home Care Organisation, Greater London
  - Participating Home Care Organisation, North West Regions
  - Participating Home Care Organisations, South West
  - Participating Home Care Organisation, West Midlands
  - Participating Home Care Organisation, Yorkshire

REFERENCES:
- [Background] Murphy J, Aryal N. Improving the provision of nutritional care for people living with dementia in care homes. Nurs Older People. 2020 Sep 22;32(5):23-29. doi: 10.7748/nop.2020.e1263. Epub 2020 Aug 12. PMID 32783432
- [Background] Murphy JL, Aburrow A, Guestini A, Brown R, Parsons E, Wallis K. Identifying older people at risk of malnutrition and treatment in the community: prevalence and concurrent validation of the Patients Association Nutrition Checklist with 'MUST'. J Hum Nutr Diet. 2020 Feb;33(1):31-37. doi: 10.1111/jhn.12710. Epub 2019 Oct 22. PMID 31637756
- [Background] Murphy JL, Holmes J, Brooks C. Nutrition and dementia care: developing an evidence-based model for nutritional care in nursing homes. BMC Geriatr. 2017 Feb 14;17(1):55. doi: 10.1186/s12877-017-0443-2. PMID 28196475
- [Derived] Yinusa G, Surr C, Thomas S, Fenge LA, Howdon D, Major J, Heward M, Taylor G, Knight H, Townson J, Murphy J. An intervention to provide nutritional care for people living with dementia at home receiving home care (TOMATO): study protocol for a single-arm feasibility study. Pilot Feasibility Stud. 2025 Nov 21;11(1):146. doi: 10.1186/s40814-025-01722-5. PMID 41272684
- See also: Project TOMATO WebPage — https://www.bournemouth.ac.uk/research/projects/tomato-nutrition-dementia-home